CLINICAL TRIAL: NCT06045312
Title: The Effect of Online Peer and Adult Education Given to Adolescents With Allergic Asthma on Their Quality of Life, Self-Efficacy, Anxiety, and Disease Knowledge and Management: A Randomized Controlled Study
Brief Title: The Effect of Online Peer and Adult Education Given to Adolescents With Allergic Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Pelin Karataş, assistant professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HF-20005
Record Dates: First submitted 2023-08-31; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Self Efficacy; Asthma; Asthma in Children
Keywords: Adolescent; Anxiety; Asthma; Knowledge; Self-efficacy; Quality of life
MeSH Terms: conditions — Asthma; Anxiety Disorders | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: In this study, there is an intervention and a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- peer education (Experimental): peer-trained group
  Interventions: Other: education
- adult education (Experimental): adult-trained group
  Interventions: Other: education
- control (No Intervention): no education

INTERVENTIONS:
Other: education — Comparison of the effectiveness of peer or adult education to adolescents with asthma
  Arms: adult education; peer education

SUMMARY:
Objectives: To examine the effect of interactive online education given by peers or adults on anxiety, self-efficacy, quality of life, and disease knowledge and management in adolescents with allergic asthma in the 10-14 age group.

Methods: The research was conducted as a randomized controlled study. The study sample consisted of 84 adolescents divided into experimental groups [receiving peer(n=28) or adult(n=28) education] and control(n=28) group. The adolescents in the peer or adults were given online interactive education concerning allergic asthma and the management thereof. The control group received only usual training.Data were collected using an Adolescent Personal Data Form, the State Anxiety Inventory for Children, the Self-Efficacy Scale for Children and Adolescents with Asthma, the Pediatric Asthma Quality of Life Questionnaire, and the Disease Knowledge and Management Questionnaire. Data were collected from the adolescents before (T0) and immediately after education (T1), and after one (T2) and three months (T3).

This study is a non-blinded randomized controlled trial. . All screened adolescents with asthma were randomly assigned to one of the three groups: the peer or adults education groups that received a 6 weeks asthma education and a control group that received usual care. The three groups were then followed prospectively immediately, 1, and 3 months after training to evaluate the effectiveness of training compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

Age was 10 to 14 years, doctor-diagnosed allergic asthma, without allergic rhinitis with a diagnosis of allergic asthma (by medical record), internet access via computer or phone, the ability to speak Turkish, willingness to participate.

Exclusion criteria were those with moderate to severe cognitive or mental health impairment and a diagnosis of allergic rhinitis in addition to the diagnosis of allergic asthma (according to medical records).

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2019-05-19 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy (SES) | 10 months
  The SES determines the degree of self-confidence of children and adolescents with asthma in taking precautions against their disease and in seeking medical assistance. This scale has 22 items. The highest possible score is 110 and the powest possible score is 22. The cut-off point score is 88. Accordingly, a score below 88 is interpreted as indicating low self-efficacy, while a score of 88 or above is interpreted as indicating high self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: pelin karataş, MsC, Principal Investigator — aydın adnan menderes universty; Hüsniye Çalışır, Study Director — aydın adnan menderes universty
Locations (1):
- Aydın Adnan Menderes University, Nursing Faculty, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No